CLINICAL TRIAL: NCT07182227
Title: A Phase 1/2 Multicenter, Open Label, Two-part Study (Single Ascending Dose [Part 1], and Dose Expansion [Part 2]) to Evaluate Safety, Tolerability and Efficacy of PS-002, a Gene Therapy for the Treatment of Adult Participants With Primary IgA Nephropathy
Brief Title: PS-002 for the Treatment of IgA Nephropathy in Adults
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Purespring Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PS-002-101; 2025-523201-14-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Immunoglobulin A (IgA) Nephropathy
Keywords: Glomerulonephritis; Nephritis; Kidney Diseases; Autoimmune Diseases; Immune System Diseases; IGA
MeSH Terms: conditions — Kidney Diseases; Glomerulonephritis; Nephritis; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Intervention Model Description: Part 1: In the dose exploration of the study, 3 different ascending dose levels will be administered using a sentinel dosing strategy Part 2: Participants will receive the optimal biological dose identified in Part 1 of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PS-002 (Experimental): Part 1: Dose escalation in three groups: Group 1: Low dose, Group 2: Intermediate Dose, Group 3: High Dose.
  Part 2: Dose expansion in a fourth group with a selected dose.
  Interventions: Genetic: PS-002

INTERVENTIONS:
Genetic: PS-002 — Adeno-associated viral vector containing the human Complement Factor I (CFI) gene

SUMMARY:
The purpose of the study is to evaluate safety, tolerability, and preliminary effectiveness following administration of PS-002 in adults with primary Immunoglobulin A (IgA) nephropathy. This will be a first-in-human study and will include participants at high risk of disease progression despite receiving current standard-of-care treatment.

Participants will be monitored for up to one year after receiving PS-002 and invited to take part in a long-term follow-up study (total follow-up: 5 years).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary IgA nephropathy (IgAN) as evidenced by renal biopsy.
* A historic kidney biopsy performed within 36 months prior to screening with reported evidence of complement component 3 (C3) deposition. If the participant had a kidney biopsy performed over 36 months prior to Screening, a new kidney biopsy should be carried out during the Screening period. This biopsy must exhibit signs of ongoing complement system activity.
* Proteinuria as assessed at the Screening visit by UPCR at least 1g/g (at least 1000 mg/g) OR total protein excretion at least 1 g/24 h (at least 1000 mg/24h) sampled from 24 h urine collection.
* eGFR calculated using the CKD-EPI formula at least 45 mL/min/1.73m^2.
* Sitting office systolic blood pressure equal to or less than 140 mmHg, diastolic blood pressure equal to or less than 90 mmHg.
* All participants must have been on best supportive care for IgAN, as per region-specific requirements defined in the protocol.

Exclusion Criteria:

* A participant has nephrotic syndrome, defined for this purpose as 24 h urine protein greater than 3.5g with concurrent hypoalbuminemia (serum albumin less than 3.0 g/dL [less than 30 g/L]).
* Any secondary IgAN defined as associated with gastrointestinal and liver disorders (liver cirrhosis, celiac disease, Crohn's disease, ulcerative colitis), autoimmune disorders (dermatitis herpetiformis, psoriasis, seronegative arthritis, systemic lupus erythematosus, rheumatoid arthritis), malignancy (IgA myeloma, lymphoma, lung cancer, renal cell cancer, cutaneous T-cell lymphoma), respiratory disorders (bronchiolitis obliterans, idiopathic pulmonary fibrosis) etc.
* Having a major concurrent non-IgAN-related disease that, in the opinion of the investigator, prevents the assessment of IgAN.
* History of malignancy; or bone marrow or organ transplant.
* History of, or currently active primary or secondary immunodeficiency, including known history of human immunodeficiency virus infection, and other severe immunodeficiency blood disorders.
* Presence of other significant medical conditions that would create an unacceptable procedure or anesthesia risk.
* Aspartate aminotransferase or alanine aminotransferase greater than 1.5 times the upper limit of normal.
* History of serious infection requiring parenteral antibiotics within the past 8 weeks prior to study drug administration.
* Participants previously treated with immunosuppressive/immunomodulatory agents such as, but not limited to, cyclophosphamide, infliximab, complement inhibitor, canakinumab, mycophenolate mofetil, mycophenolate sodium, cyclosporine, tacrolimus, everolimus, or systemic corticosteroids (exposure greater than 7.5mg/day prednisone/prednisolone equivalent) within 90 days (or 180 days for rituximab) prior to Screening. Participants previously or currently receiving oral budesonide (Kinpeygo/Tarpeyo) require wash out for 90 days prior to the study drug administration.
* Exposed to a live or attenuated vaccine within the 6 weeks prior to study drug administration.
* Participants with a known sensitivity or intolerance to corticosteroid therapy.
* Known hypersensitivity to study drug ingredients.
* Prior treatment with PS-002 or any other gene therapy, or participation in any other investigational trial during this study.
* Positive serology for hepatitis B or C, i.e., positive hepatitis B surface antigen or hepatitis C ribonucleic acid (RNA) viral load positive.
* Participants treated with potentially hepatotoxic medications unless they have been monitored in accordance with the drug label and have received a stable dose since >90 days prior to dosing without clinically significant liver enzyme fluctuations.

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with: Treatment-Emergent Adverse Events (TEAEs) and serious TEAEs, TEAEs and serious TEAEs related to PS-002, TEAEs and serious TEAEs related to the PS-002 administration procedure | Screening up to Week 48

SECONDARY OUTCOMES:
Change in proteinuria as measured by Urine Protein:Creatinine Ratio (UPCR) derived from 24 hr urine collection | Baseline to Week 36
Change from baseline in proteinuria as measured by urine protein creatinine ratio (UPCR) from spot urine collection. [UPCR (g/g) will be calculated from spot urine collection (first morning void)] | Baseline to Week 48
Change from baseline in proteinuria as measured by urine albumin:creatinine ratio (UACR). [UACR (g/g) will be calculated from spot urine collection (first morning void)] | Baseline to Week 48
Change from baseline in proteinuria as measured by UACR from 24 hour urine collection. [UACR (mg/day) will be calculated from 24 hour urine collection at Week 36 only] | Baseline to Week 36
Change from baseline in creatinine and estimated Glomerular Filtration Rate (eGFR) values calculated using the Chronic Kidney Disease Epidemiology (CKD-EPI) creatinine formula | Baseline to Week 48
Change from baseline in urinary soluble terminal complement complex (sC5b-9) levels | Baseline to Week 48
Time to worsening of kidney function. Defined as: 1) sustained eGFR decline by at least 40 percent, 2) onset of end-stage kidney disease, 3) initiation of renal replacement therapy, or 4) all-cause mortality | Baseline to Week 48

CONTACTS AND LOCATIONS:
Locations (11):
- United States (3):
  - University of Miami Hospital, Miami, Florida
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan Hospital, Ann Arbor, Michigan
- United Kingdom (8):
  - Manchester University NHS Foundation Trust, Manchester, Greater Manchester
  - Salford Royal Hospital, Northern Care Alliance NHS Foundation Trust, Manchester, Greater Manchester
  - Leicester General Hospital, Leicester, Leicestershire
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - Southmead Hospital, Bristol
  - Cardiff and Vale University Health Board, Cardiff
  - Royal Infirmary of Edinburgh Clinical Research Facility, Edinburgh
  - The Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: No
IPD data are not planned to be shared at this time due to patient privacy concerns with consideration of the small sample size for this open-label study